CLINICAL TRIAL: NCT03915535
Title: Impact of Two Formulations of Fish Oil Monoglycerides on the Modulation of Mitochondrial Functions and Lactate Threshold in Athletes. A Pilot Study
Brief Title: Impact of Fish Oil Monoglycerides on the Modulation of Mitochondrial Functions and Lactate Threshold
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Several impacts of COVID-19 on recruitment and organization
Sponsor: Samuel Fortin (Industry)
Responsible Party: Sponsor-Investigator, Samuel Fortin, Principal Investigator, SCF Pharma
Organization: SCF Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PSP-MG01
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Healthy Athletes
MeSH Terms: interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; 1-eicosapentaenoylglycerol

STUDY DESIGN:
Intervention Model Description: This is a two parallel groups study without randomisation.12 subjects will be enrolled in group A. Afterwards, the remaining 12 subjects will be enrolled in group B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaxSimil (Active Comparator): Subjects of group A will receive a constant daily dose of 4.3g of MaxSimil, a combination of EPA + DHA in proportions of 500/200, for a period of 90 days.
  Interventions: Dietary Supplement: Eicosapentaenoic acid + Docosahexaenoic acid
- MAG-EPA (Experimental): Subjects of group B will receive a constant daily dose of 4.4g of MAG-EPA, a purified formulation of EPA with traces of DHA (730/050), for a period of 90 days.
  Interventions: Dietary Supplement: Eicosapentaenoic acid

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid + Docosahexaenoic acid — Monoglyceride Omega-3 fish oils
  Other Names: MaxSimil
  Arms: MaxSimil
Dietary Supplement: Eicosapentaenoic acid — Monoglyceride Omega-3 fish oil
  Other Names: MAG-EPA
  Arms: MAG-EPA

SUMMARY:
he objective of this study is to compare the effects two different formulations of fish oil monoglycerides on the mitochondrial functions and on the lactate threshold of athletes during a high intensity exercise. Twenty four (24) subjects will be enrolled in the study and followed for a period of 90 days. A first visit will capture all the baseline parameters and will be followed by two subsequent visits (at day 45 and at day 90) where the same measurements will be done. The subjects will be divided in two parallel groups. Subjects of group A will receive a constant daily dose of 4,3g eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA) whereas subjects of group B will receive a constant daily dose of 4,4g of EPA only. Subjects will be treated from day 1 to day 90 without interruption or modification to their regimen.

DETAILED DESCRIPTION:
Twenty four (24) subjects will be enrolled and sequentially assigned to one of the two parallel treatment formulations. The study population will be men and women of 19 years and older with no allergy or history of allergy to fish. Participants must practice at least 6 hours of intense physical activity per week as a life habit and must not have taken omega-3 monoglycerides within the last 30 day prior to study enrollment. Pregnant or lactating women will be excluded from the study.

The objective of this study is to compare the effects of MaxSimil, a combination of EPA and DHA monoglycerides with the monoglyceride EPA alone (MAG-EPA). For each group, the primary objectives will be to measure the changes in mitochondrial functions (LEAK, RCR and OKPHOS) and in the lactate threshold of athletes throughout the study. The program is similar for each visit and contains: fasting bood draw, standardized breakfast, health questionnaire, vital signs and the lactate threshold test. The latter consists of a standardized exercise on a stationary bike during which the blood lactate concentration as well as blood sugar concentration will be monitored by capillary puncture at determined time intervals. The fasting blood draw will be used for the analysis of mitochondrial functions, the omega-3 index as well as the quantification of cytokines such as Interleukine-1, Interleukine-6 and the C-reactive protein (CRP). All the data collected after 45 and 90 days will be compared to the baseline measurements.

The screening tasks include pregnancy testing for women, collection of demographic information and baseline health/ life habits questionnaire.

Study Medication will be dispensed to subjects at visit 1. Medication will be self-administered by the subjects at home. Subjects will be given a diary to fill-out in case of missed doses, concomitant medication intake, adverse events or significant changes in life habits.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged of at least 19 years old.
* Availability for the entire duration of the study and willingness to participate based on the information provided in the Informed Consent Form (ICF) duly read and signed by the latter.
* Participant with no intellectual problems that may limit the validity of consent to participate in the study or the compliance with the protocol requirements, ability to cooperate adequately, to understand and to observe the instructions of the physician or designee.
* Participant having no difficulty swallowing tablets or capsules.
* Participant who engages in at least six hours of physical activity (intense sport training) per week.

Exclusion Criteria:

* Allergy to fish or history of allergic reactions attributable to fish or to a fish oil-like compound.
* Female who are pregnant or are lactating.
* Intake of omega-3 monoglycerides in the 30 days prior to day 1 of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Quantification of mitochondrial functions (Oxphos. Leak, RCR) | 90 days per subject. About seven months for the whole study.
  For both group, mitochondrial functions will be measured at baseline, after 45 days and after 90 days of treatment. Potential improvement will be compared between groups
Measurement of the improvement of the Lactate threshold in athletes | 90 days per subject. About seven months for the whole study.
  For both group, lactate threshold will be measured at baseline, after 45 days and after 90 days of treatment. Potential improvement will be compared between groups

SECONDARY OUTCOMES:
Quantification of inflammation markers (Cytokines) | 90 days per subject. About seven months for the whole study.
  At each visit ( V1 = baseline, V2 = day 45, V3 = day 90), a blood sample will be taken to quantify the following cytokines: Interleukine-1, Interleukine-6 and C-reactive Protein. Inflammation markers such as cytokines might be indicators of good responders to Omega-3 treatments & prevention.
measurement of the Omega-3 index | 90 days per subject. About seven months for the whole study.
  At each visit ( V1 = baseline, V2 = day 45, V3 = day 90), a blood sample will be taken to measure the omega-3 index (total amount of EPA + DHA in the red blood cells). This parameter helps to monitor the subject's exposition to treatment.
Recording and monitoring of life habits | 90 days per subject. About seven months for the whole study.
  At each visit ( V1 = baseline, V2 = day 45, V3 = day 90), subjects will be questioned about their life habits such as: smoking, alcohol intake, number of fish meals per week, sports habits, vitamins and dietary supplements intake. These informations should help to control bias in primary objectives response and give further hints to what makes good responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Santé 2000, Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No